CLINICAL TRIAL: NCT01265888
Title: A Phase 2, Open-Label, Dose-Escalation Study in Subjects With Pulmonary Arterial Hypertension, (PAH, WHO Group 1) and Pulmonary Hypertension Secondary to Idiopathic Pulmonary Fibrosis, (PH-IPF WHO Group 3) Using Inhaled GeNOsyl.
Brief Title: Study in Subjects With PAH and PH Secondary to IPF Using Inhaled GeNOsyl.
Acronym: PHiano
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Geno LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol # GeNO-P-2010-002; PHiano (Other: Study Sponsor (GeNO, LLC))
Record Dates: First submitted 2010-12-20; First posted 2010-12-23 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Pulmonary Arterial Hypertension; Idiopathic Pulmonary Fibrosis
Keywords: PAH; PH IPF
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dosing Group 1 (Experimental): 1 Liter per Minute (LPM)of inhaled nitric oxide via nasal cannula: approximately 5 parts per million (ppm)
  Interventions: Drug: Inhaled Nitric Oxide
- Dosing Group 2 (Experimental): 2 LPM of inhaled nitric oxide via nasal cannula: approximately 15 ppm
  Interventions: Drug: Inhaled Nitric Oxide
- Dosing Group 3 (Experimental): 4 LPM of inhaled nitric oxide via nasal cannula: approximately 20 ppm
  Interventions: Drug: Inhaled Nitric Oxide

INTERVENTIONS:
Drug: Inhaled Nitric Oxide — Inhaled nitric oxide 80 ppm via nasal cannula at 1 LPM for 15 minutes followed by placebo washout of 15 minutes inhalation of medical grade air (or prescribed supplemental oxygen), and then inhaled nitric oxide 80 ppm via nasal cannula at 1 LPM
  Other Names: GeNOsyl
  Arms: Dosing Group 1
Drug: Inhaled Nitric Oxide — Inhaled nitric oxide 80 ppm via nasal cannula at 1 LPM for 15 minutes followed by placebo washout of 15 minutes inhalation of medical grade air (or prescribed supplemental oxygen), and then inhaled nitric oxide 80 ppm via nasal cannula at 2 LPM
  Other Names: GeNOsyl
  Arms: Dosing Group 2
Drug: Inhaled Nitric Oxide — Inhaled nitric oxide 80 ppm via nasal cannula at 1 LPM for 15 minutes followed by placebo washout of 15 minutes inhalation of medical grade air (or prescribed supplemental oxygen), and then inhaled nitric oxide 80 ppm via nasal cannula at 4 LPM
  Other Names: GeNOsyl
  Arms: Dosing Group 3

SUMMARY:
A Phase 2 open label, dose escalation study to find the minimally and maximum effective dose (dose beyond which no further effect on PVR is seen) of inhaled nitric oxide generated by the GeNOsyl® System compared to placebo.

DETAILED DESCRIPTION:
Up to 54 subjects undergoing RHC are planned in this study, and shall include subjects meeting eligibility criteria classified as WHO Group 1 PAH or WHO Group 3 IPF-PH. Subjects will receive inhaled nitric oxide from the GeNOsyl® System to characterize the hemodynamic response and evaluate safety and tolerability.

Dose cohorts of approximately 5, 15, and 20 ppm nitric oxide in air will be studied. Different dose levels will be achieved by varying the flow rate of the drug substance (80 ppm NO2 in balance air) delivered to the subject via nasal cannula. Each subject will receive two different doses of inhaled nitric oxide separated by a placebo (medical grade air or supplemental oxygen) washout. Eligible subjects will be assigned to a dosing cohort in an escalating manner to receive study drug (80 ppm nitric oxide in air.)

ELIGIBILITY:
INCLUSION CRITERIA:

PAH and PH-IPF

* WHO Functional Class (or equivalent classification) II - IV.
* Subjects using supplemental oxygen must be receiving a stable course of therapy for a minimum of 14 days prior to study drug administration.
* All subjects' oxygen saturation must be > or = to 88% at time of treatment
* Echocardiogram within 6 months of baseline showing no signs of clinically significant left sided heart disease
* Females of child-bearing potential with a negative urine pregnancy test, or a documented surgical sterilization, or is post-menopausal prior to administration of investigational product. Females of childbearing potential must be practicing adequate birth control.

PAH (WHO Group 1) ONLY-Inclusion

* Documented diagnosis of WHO Group 1 PAH, (limited to, idiopathic, heritable, drug and toxin induced, associated with connective tissue disease, portal hypertension, repaired congenital heart disease, HIV); documented by a previous RHC and hemodynamics consistent with PAH, WHO Group 1
* Pulmonary Function Testing within 6 months prior to screening/enrollment shows no evidence of interstitial lung disease (TLC<70%) or obstructive lung disease (FEV1/FVC ratio <50%)
* Receiving a stable course of approved PAH oral mono therapies for a minimum of 14 days prior to treatment period
* Must be 18-80 year of age

PH-IPF (WHO Group 3) ONLY-Inclusion

* Documented diagnosis of probable or definite IPF using ATS/ERS criteria
* Previous transbronchial biopsy, if performed, shows no features to support a definitive alternative diagnosis
* Previous bronchoalveolar lavage, if performed, shows no features that provides an alternative diagnosis
* FVC > or = 40% within 6 months of baseline visit
* Diagnosis of PH based on hemodynamic requirements
* Age 40-85.
* Diagnosis of IPF > or = 3 months prior to study drug administration
* Diagnosis of PH based on the following hemodynamic criteria (PAPm > or = 25 mmHg (at rest) / PCWP or LVED < or =15 mmHg and / PVR >3 Wood Units)

EXCLUSION CRITERIA:

PAH and PH-IPF

* Have any other disease associated with pulmonary hypertension (i.e. Group II, IV or V).
* Documented uncontrolled systemic hypertension.
* Left ventricular ejection fraction (LVEF) < 40%.
* Have chronic kidney disease stage IV or worse, or requires dialysis.
* Be receiving an investigational drug, have in place an investigational device, or have participated in an investigational drug study within past 30 days.
* Have had an atrial septostomy.
* Have anemia or any other ongoing condition that would interfere with the interpretation of study assessments.
* Have any serious or life-threatening disease other than conditions associated with PAH or PH-IPF (e.g. malignancy requiring aggressive chemotherapy, renal dialysis, etc.)
* Significant, ongoing alcohol or drug abuse, or unstable psychiatric status.
* Receiving inhaled or parenteral prostacyclins or a non-approved combination of approved oral PAH therapy.
* Pregnant or lactating subjects

PAH (WHO Group 1) ONLY-Exclusion

* Have had any changes to chronic therapy (including but not limited to oxygen, a different category of vasodilator, a diuretic, digoxin) for PAH added within 14 days of study drug administration. Anticoagulants are allowed to be discontinued per institutional standard of care.
* History of untreated sleep apnea within three months of study drug administration.
* History of hemodynamically significant left-sided heart disease or evidence of left-sided heart disease.

PH-IPF (WHO Group 3) ONLY-Exclusion

* Diagnosis of PH primarily due to etiology other than IPF.
* FEV/FVC ratio < 60% documented within 6 months of baseline visit.
* Hospitalization for acute exacerbation of IPF within 30 days of baseline visit.
* Recent active pulmonary or upper respiratory tract infection.
* Receiving any approved PAH therapy within 30 days of study drug administration.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Identify the minimally and maximum effective doses of inhaled nitric oxide generated by the GeNOsyl® System compared to placebo. | through end of Right Heart Catheterization procedure (Treatment Phase approximately 3 hours)
  Assess mean change in pulmonary vascular resistance (PVR) for study drug dose 2 compared to placebo.
  Assess change from pre-dose to end-of-hemodynamic assessment for study drug dose 1.
  Assess change from placebo to end-of-hemodynamic assessment for study drug dose 2.

SECONDARY OUTCOMES:
Assess the safety and tolerability of nitric oxide generated by the GeNOsyl® System in subjects with WHO Group 1 PAH and WHO Group 3 PH-IPF. | through end of study (approximately 30 days after treatment visit)
Evaluate the pharmacokinetics of total nitrates/nitrites and methemoglobin produced following inhalation of nitric oxide via the GeNOsyl® System. | up through 24 hrs after treatment period for subjects participating in PK sub-study
  Individual pharmacokinetic parameters for total nitrates/nitrites and methemoglobin will be summarized with descriptive characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Suplick, Study Director — Geno LLC
Locations (10):
- United States (10):
  - University of Alabama @ Birmingham, Birmingham, Alabama
  - VA Greater LA Health Care System-UCLA, Los Angeles, California
  - University of California- Davis Medical Center, Sacramento, California
  - National Jewish Health, Denver, Colorado
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - Washington University School of Medicine, St Louis, Missouri
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - Ohio State University, Martha Morehouse Medical Plaza, Columbus, Ohio
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes